CLINICAL TRIAL: NCT00760006
Title: Efficacy of Preoperative Prophylactic Antibiotics in Preventing Complications in the Primary Repair of Cleft Palates
Brief Title: Preventing Complications in Cleft Palate Repair With Antibiotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Losee (Other)
Responsible Party: Sponsor-Investigator, Joseph Losee, Ross H. Musgrave Professor of Pediatric Plastic Surgery Executive Vice-Chair and Program Director Department of Plastic Surgery University of Pittsburgh Medical Center, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07090352
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Cleft Palates
Keywords: cleft secondary palate; primary closure of secondary cleft palate; Prophylactic Antibiotics; Unasyn; Cleft Palate
MeSH Terms: conditions — Cleft Palate | interventions — sultamicillin; Ampicillin; Sulbactam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unasyn Antibiotic Arm (Active Comparator): Unasyn® is a parenteral antibiotic that combines ampicillin with sulbactam, a beta-lactamase inhibitor. All subjects enrolled in the study will receive a single dose of antibiotic or saline solution (placebo control) intravenously, as the IV will already be in place as standard of care for surgery. The study aims to assess the efficacy of the prophylactic antibiotic in cleft surgery to: decrease the incidence of surgical site infections, speed the progression of postoperative healing, improve the final quality of wound healing achieved, and decrease the rate of palatal fistula formation.
  Interventions: Drug: Unasyn
- Saline Placebo Arm (Placebo Comparator): Saline Placebo. All subjects enrolled in the study will receive a single dose of antibiotic or saline solution (placebo control) intravenously, as the IV will already be in place as standard of care for surgery. This will act as the placebo control.
  Interventions: Other: saline solution

INTERVENTIONS:
Drug: Unasyn — Subjects will receive the antibiotic or the saline placebo 30 minutes prior to the initial incision in their palatoplasty procedure. The FDA approved antibiotic used for this study is Unasyn. Unasyn is a first-line measure, used by ENT surgeons at Children's Hospital of Pittsburgh for antibiotic treatment of virtually all ear, nose and throat infections. The use of Unasyn for this study is off-label as with the majority of antibiotics used with children. Subjects will receive a one time dose of 50mg/kg prior to surgery, not to exceed a total of 2gm
  Other Names: ampicillin; sulbactam
  Arms: Unasyn Antibiotic Arm
Other: saline solution — Subjects will receive a one time dose of 50mg/kg prior to surgery, not to exceed a total of 2gm.
  Other Names: Salt solution
  Arms: Saline Placebo Arm

SUMMARY:
The primary objective of this study is to determine the efficacy of administering a single dose of preoperative antibiotics to prevent complications in patients undergoing primary closure of a cleft secondary palate. Secondary objective of this study is to evaluate the effects of preoperative antibiotics administered on post operative outcome following primary closure of cleft secondary palate. The study aims to assess the efficacy of prophylactic antibiotics in cleft surgery to

* decrease the incidence of surgical sight infections
* speed the progression of postoperative healing
* improve the final quality of wound healing achieved
* decrease the rate of palatal fistula formation

DETAILED DESCRIPTION:
During the initial clinical visit, the clinical diagnosis of a cleft secondary palate or submucous cleft will be made. Other associated clinical findings such as unilateral/bilateral cleft lip, unilateral/bilateral cleft primary palate, Veau cleft palate classification, and associated syndromic diagnosis will be recorded. The severity of the cleft palate will be documented by measuring the width of the cleft and the hard-soft palate juncture. The patients will proceed through the standardized cleft treatment protocol as mandated by their specific anatomic findings. These include possible naso-alveolar molding, lip-adhesion procedures, and cleft lip repair procedures. The patients will be followed regularly in clinic and will undergo a palatoplasty procedure to repair their cleft secondary palate when clinically indicated, typically between the age of 9 and 14 months. Patients who present for treatment late will be operated on when clinically appropriate, as determined by the plastic surgeon. A Furlow palatoplasty procedure is the typical palatoplasty procedure performed by the primary investigator, but other procedures such a Von Langenbeck pushback palatoplasty may be performed as dictated by the clinical scenario.

Subjects will be randomized via aid from statisticians in the Clinical and Translational Science Institute (CTSI) here at the University of Pittsburgh. This will enable the research pharmacist at Children's Hospital of Pittsburgh, to send either the antibiotic or the saline placebo to the operating room in a blinded manner. All subjects enrolled in the study will receive a single dose of antibiotic or saline solution (placebo control) intravenously, as the IV will already be in place as standard of card for surgery. Subjects will receive the antibiotic or the saline placebo 30 minutes prior to the initial incision in their palatoplasty procedure. The FDA approved antibiotic used for this study is Unasyn. Unasyn is a first-line measure, used by ENT surgeons at Children's Hospital of Pittsburgh for antibiotic treatment of virtually all ear, nose and throat infections. The use of Unasyn for this study is off-label as with the majority of antibiotics used with children. Subjects will receive a one time dose of 50mg/kg prior to surgery, not to exceed a total of 2gm. This constitutes the focus of the study, and is the only variation from standard treatment.

Patients will be admitted to the hospital, and will be discharged home when they are in no respiratory distress, have adequate pain control, and are able to tolerate adequate PO intake. This is generally on post-operative day 2. All patients will be prescribed pain medications. Parents will be provided with, and counseled how to properly use arm splints for 14 days postoperatively. They will also be taught how to feed the child with syringe feeds. These measures prevent the child from traumatizing the suture lines with bottles, hands and foreign bodies.

Screening procedures will consist of a medical history and physical examination by a Pediatric Plastic Surgeon to determine what type of cleft palate repair is necessary. This is the same standard exam and medical/surgical work-up that any patient would receive if they were treated by the Cleft-Craniofacial Clinic in Children's Hospital of Pittsburgh of UPMC and not enrolled in this study. This aspect of care will not vary from routine treatment. All patients will be seen in weekly postoperative follow-up in the Cleft-Craniofacial Center. Documentation of these postoperative visits will include notation of signs of surgical sight infections, such as continued fevers, erythema, swelling, discharge, dehiscence, pain, and the presence of nonviable tissue. The progression of wound healing will be quantified on a scale of 1 to 4. Wounds will be classified as Stage 1 healing when there is complete union of the mucosa, and no irregularities or separation. Stage 2 healing will be documented for wounds with minor incisional irregularities or incomplete healing. Stage 3 healing will be documented when the wound exhibits worrisome mucosal viability, partial dehiscence of the oral mucosal closure, erythema, purulent drainage, or exposure of the alloderm patch. Stage 4 healing will include patients with a palatal fistula. Any patients with clinical signs and symptoms of thrush, a fungal infection of the mouth and esophagus, will have cultures of the lesions sent to confirm the diagnosis. These patients will be immediately started on a seven day course of oral fluconazole, with an initial dose of 6mg/kg, followed by daily dose of 3mg/kg, as recommended by Dr. Andrew Nowalk, MD. Patients will be seen in clinic weekly until they have reached stage 1 healing, or until the presence of a palatal fistula is documented. We anticipate a minimum of less than 2 months to a maximum of 1 year for follow-up will be necessary to document either stage 1 healing or the presence of a palatal fistula in nearly all cases. The primary endpoints measured will be 1) the incidence of surgical sight infections, 2) the incidence of palatal fistula 3) the average time needed to achieve stage 1 healing, 4) the incidence of cases with healing delayed more than one standard deviation from the average, 5) the incidence of thrush, a fungal infection of the mouth and esophagus, and 6) the incidence of allergic/drug reactions to the study drug. Surveillance for other factors such as hospital length of stay, postoperative bleeding events, postoperative respiratory distress, and diagnosis of a sepsis will be recorded as secondary endpoints.

Data collection will include patient characteristics such as, but not limited to, Veau cleft classification, width of the cleft defect, presence of associated cleft lip or primary palate, presence of syndromic diagnosis, and use of alloderm for repair augmentation, and the administration of intraoperative steroids. The two study groups will be compared on the basis of these characteristics to determine if statistically significant differences exist between the two groups. Endpoint data will be collected as discussed above, and the outcomes for the placebo and antibiotic group will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as having cleft palates undergoing palatoplasty between the ages of 3 months and 18 years will be included in this study. Palatoplasty is the current standard of care in the sequence of treatment for cleft secondary palates. Pediatric plastic surgeons work primarily with children, and have undergone extensive training during their residencies and pediatric surgical fellowships to do so. Children will be evaluated initially at the Cleft-Craniofacial Center at the Children's Hospital of Pittsburgh of UPMC, which is set up to accommodate children of all ages and their families. Approximately 300 children will be required to contribute to a meaningful analysis.

Exclusion Criteria:

* All patients requiring prophylactic antibiotics for spontaneous bacterial endocarditis, with documented allergic reactions to the ampicillin-sulbactam, and with known immunodeficiencies or immunodeficiency associated syndromes, such as the 22q chromosomal deletion, will be excluded from study participation.
* Selection will be based on the parent's willingness to allow their child to participate in the study.
* Children already receiving antibiotics at the time of their surgery will be evaluated distinctly, though they will not be included in the antibiotic or the placebo groups

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 224 (Actual)
Dates: Start 2008-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Losee, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Improved national prevalence estimates for 18 selected major birth defects--United States, 1999-2001. MMWR Morb Mortal Wkly Rep. 2006 Jan 6;54(51):1301-5. PMID 16397457
- [Background] Chuo CB, Timmons MJ. The bacteriology of children before primary cleft lip and palate surgery. Cleft Palate Craniofac J. 2005 May;42(3):272-6. doi: 10.1597/03-108.1. PMID 15865461
- [Background] Mercer NS. The use of preoperative swabs in cleft lip and palate repair. Br J Plast Surg. 2002 Mar;55(2):176-7. doi: 10.1054/bjps.2001.3776. No abstract available. PMID 11987971
- [Background] JOLLEYS A, SAVAGE JP. Healaing defects in cleft palate surgery--the role of infection. Br J Plast Surg. 1963 Apr;16:134-9. doi: 10.1016/s0007-1226(63)80094-6. No abstract available. PMID 13957936
- [Background] JACKSON DM, LOWBURY EJ, TOPLEY E. Chemotherapy of Streptococcus pyogenes infection of burns. Lancet. 1951 Oct 20;2(6686):705-11. doi: 10.1016/s0140-6736(51)91478-x. No abstract available. PMID 14874485
- [Background] McClelland RMA, Patterson TJS. The influence of penicillin on the complication rate after repair of clefts of the lip and palate. Br J Plast Surg. 1963; 16:144-145
- [Background] Marzoni FA, Kelly DR. Bacteremia following cleft palate repair--a prospective study. Ann Plast Surg. 1983 Jun;10(6):473-4. doi: 10.1097/00000637-198306000-00006. PMID 6881863
- [Background] Crawford JJ, Fischer ND. Oral and respiratory flora of individuals with normal and repaired palatal clefts. Cleft Palate J. 1971 Apr;8:166-76. No abstract available. PMID 5283309

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol exclusion criteria includes children already receiving antibiotics at the time of their surgery, and will be evaluated distinctly, but will not be included in the antibiotic or placebo groups. Therefore, only participants receiving preoperative antibiotics are considered for our outcome measure.
Groups:
- Unasyn Antibiotic Arm: Active Comparator: Unasyn® is a parenteral antibiotic that combines ampicillin with sulbactam, a beta-lactamase inhibitor. All subjects enrolled in the study will receive a single dose of antibiotic or saline solution (placebo control) intravenously, as the IV will already be in place as standard of care for surgery. The study aims to assess the efficacy of the prophylactic antibiotic in cleft surgery to: decrease the incidence of surgical site infections, speed the progression of postoperative healing, improve the final quality of wound healing achieved, and decrease the rate of palatal fistula formation.
  Subjects will receive the antibiotic or the saline placebo 30 minutes prior to the initial incision in their palatoplasty procedure.
  Subjects will receive a one time dose of 50mg/kg prior to surgery, not to exceed a total of 2gm
- Saline Placebo Arm: Other Names:
  * Salt solution
  * Saline Solution Subjects will receive the antibiotic or the saline placebo 30 minutes prior to the initial incision in their palatoplasty procedure.
  Subjects will receive a one time dose of 50mg/kg prior to surgery, not to exceed a total of 2gm
Period: Overall Study
Arm/Group | Unasyn Antibiotic Arm | Saline Placebo Arm
Started | 86 | 138
Completed | 86 | 138
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Unasyn Antibiotic Arm: Unasyn® is a parenteral antibiotic that combines ampicillin with sulbactam, a beta-lactamase inhibitor. All subjects enrolled in the study will receive a single dose of antibiotic or saline solution (placebo control) intravenously, as the IV will already be in place as standard of care for surgery. The study aims to assess the efficacy of the prophylactic antibiotic in cleft surgery to: decrease the incidence of surgical site infections, speed the progression of postoperative healing, improve the final quality of wound healing achieved, and decrease the rate of palatal fistula formation.
  Subjects will receive the antibiotic or the saline placebo 30 minutes prior to the initial incision in their palatoplasty procedure.
  Subjects will receive a one time dose of 50mg/kg prior to surgery, not to exceed a total of 2gm
- Total: Total of all reporting groups
Arm/Group | Unasyn Antibiotic Arm | Saline Placebo Arm | Total
Number analyzed (Participants) | 86 | 138 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86 | 138 | 224
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 62 | 101
  Male | 47 | 76 | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 138 | 224

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fistula or Delayed Wound Healing Following Palatoplasty
Description: Primary outcomes of fistula or delayed wound healing following palatoplasty were measured in two groups of patients. This outcome measure addresses both objectives noted in the summary of the study description.
Time Frame: We anticipate a minimum of less than 2 months to a maximum of 1 year for follow-up will be necessary to document either stage 1 healing or the presence of a palatal fistula in nearly all cases.
Population: Only participants receiving preoperative antibiotics are considered for this outcome measure. Please refer to the exclusion criteria listed in the initial protocol -- "Children already receiving antibiotics at the time of their surgery will be evaluated distinctly, though they will not be included in the antibiotic or placebo groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Unasyn Antibiotic Arm | Saline Placebo Arm
Number analyzed (Participants) | 86 | 138
Participants
  Fistula | 3 | 2
  Delayed Wound Healing | 18 | 21

ADVERSE EVENTS:
Description: As noted in the protocol exclusion criteria, children already receiving antibiotics at the time of their surgery were evaluated distinctly, though they were not included in the antibiotic or placebo groups. Only participants receiving preoperative antibiotics are considered for outcome measure and adverse events.
Arm/Group | Unasyn Antibiotic Arm | Saline Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/138
Other Adverse Events (participants affected / at risk) | 0/86 | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes